CLINICAL TRIAL: NCT02503722
Title: A Phase 1 Trial of MLN0128 (TAK-228) in Combination With Osimertinib (AZD9291) in Advanced EGFR Mutation Positive Non-Small Cell Lung Cancer (NSCLC) After Progression on a Previous EGFR Tyrosine Kinase Inhibitor
Brief Title: Testing the Combination of MLN0128 (TAK-228) and AZD9291 in Advanced EGFR (Epidermal Growth Factor Receptor) Mutation Positive Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01139; NCI-2015-01139 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PJC-020; 9910/PJC-020; 9910 (Other: University Health Network Princess Margaret Cancer Center LAO); 9910 (Other: CTEP); UM1CA186644 (NIH); UM1CA186689 (NIH)
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage III Lung Non-Small Cell Cancer AJCC v7; Stage IIIA Lung Non-Small Cell Cancer AJCC v7; Stage IIIB Lung Non-Small Cell Cancer AJCC v7; Stage IV Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sapanisertib, osimertinib) (Experimental): Patients receive sapanisertib PO QD on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26 (day 1 is omitted in cycle 1). Patients also receive osimertinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Osimertinib; Other: Pharmacological Study; Drug: Sapanisertib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Osimertinib — Given PO
  Other Names: AZD 9291; AZD-9291; AZD9291; Mereletinib
Other: Pharmacological Study — Correlative studies
Drug: Sapanisertib — Given PO
  Other Names: INK-128; INK128; MLN-0128; MLN0128; TAK-228

SUMMARY:
This phase I trial studies the side effects and best dose of sapanisertib when given together with osimertinib in treating patients with stage IV EGFR mutation positive non-small cell lung cancer that has progressed after treatment with an EGFR tyrosine kinase inhibitor. Sapanisertib and osimertinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and recommended phase II dose (RP2D) of sapanisertib (MLN0128) (TAK-228) in combination with osimertinib (AZD9291) in patients with advanced epidermal growth factor receptor mutation positive (EGFRm) non-small cell lung cancer (NSCLC) and who are resistant to previous EGFR-tyrosine kinase inhibitor (TKI) therapy. (Dose escalation phase) II. To evaluate the safety and preliminary efficacy of MLN0128 (TAK-228) in combination with osimertinib (AZD9291) in patients with advanced EGFRm NSCLC who are resistant to previous EGFR-TKI therapy with first line osimertinib. (Dose expansion phase)

SECONDARY OBJECTIVES:

I. To evaluate pharmacokinetic profiles of MLN0128 (TAK-228) in combination with osimertinib (AZD9291).

II. To evaluate the response rate, disease control rate and progression free survival of the combination.

III. To explore biomarkers of response and resistance to the combination by studying baseline biopsies, resistance biopsies, and serial plasma deoxyribonucleic acid (DNA) specimens.

OUTLINE: This is a dose-escalation study of sapanisertib.

Patients receive sapanisertib orally (PO) once daily (QD) on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26 (day 1 is omitted in cycle 1). Patients also receive osimertinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and then every 8 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IV or recurrent/metastatic histologically or cytologically confirmed non-squamous NSCLC
* NSCLC must harbor an EGFR activating mutation (Exon 21 L858R, Exon 19 deletion)
* Progressive disease on osimertinib (AZD9291) given first line
* For the dose expansion portion ONLY, patient must: 1) have progression of disease with first line osimertinib administered for advanced or metastatic disease as the last previous systemic treatment, 2) be treatment naïve for other 3rd generation EGFR-TKI (CO-1686) and mTOR inhibitors
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, defined as at least one lesion that can be accurately measured in at least one dimension >= 10 mm (>= 1 cm) by computed tomography (CT) imaging or magnetic resonance imaging (MRI) within 28 days prior to start of protocol therapy; the CT from a combined positron emission tomography (PET)/CT may be used if it is of diagnostic quality; laboratory parameters are not acceptable as the only evidence of disease
* For the dose expansion, no other systemic therapies for advanced/metastatic disease is permissible after first line osimertinib
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Patients with a prior history of brain metastases are eligible provided:

  * The brain metastases have been treated; patients with small brain metastases for which radiation or surgery is not indicated, may be eligible on discussion with the study chair. Brain metastases that were managed with first line osimertinib is permissible, provided that the brain metastases are stable on a baseline MRI and for whom radiation or surgical resection is not indicated
  * The patient is asymptomatic from the brain metastases
  * Corticosteroids and anti-epileptic drugs prescribed for the management of brain metastases have been discontinued at least 7 days prior to registration
  * The brain metastases are stable on pre-registration imaging
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin >= 90 g/L (or >= 9 g/dL)
* Platelets >= 100 x 10^9/L
* Calculated creatinine clearance of > 50 mL/min using Cockcroft Gault equation or 24-hour urine sampling
* Total bilirubin =< 1.5 institutional upper limit of normal
* Aspartate transaminase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Fasting plasma glucose =< 130 mg/dL (or 7.2 mmol/L)
* Glycosylated hemoglobin (Hb A1c) =< 7.0%
* Fasting triglycerides =< 300 mg/dL (3.42 mmol/L)
* Cholesterol =< 300 mg/dL (7.75 mmol/L)
* Fridericia's correction formula (QTcF) =< 470 msec
* Patients must have had sufficient time between a prior therapy and resolution of toxicities from the prior therapies prior to registration as follows:

  * Prior EGFR inhibitor: A minimum of 7 days must have elapsed from the last dose of the prior EGFR inhibitor and resolution of any drug-related toxicity to =< grade 1 except for alopecia
  * Chemotherapy: A minimum of 21 days must have elapsed from the last dose and resolution of toxicity to =< grade 1 excluding =< grade 2 peripheral neuropathy or alopecia
  * Surgery: A minimum of 21 days must have elapsed following major surgery and resolution of toxicity to < grade 1 and complete wound healing must have occurred
  * Radiation: A minimum of 14 days must have elapsed following radiation therapy and resolution of all radiation induced toxicity excluding alopecia
  * Treatment with an investigational drug: A minimum of 3 months or five half-lives of the compound, whichever is greater, must have elapsed from last treatment date
* Ability to understand and the willingness to sign a written informed consent document
* Available for follow-up of their disease after treatment until progressive disease is documented and resolution of related adverse events until < grade 2

Exclusion Criteria:

* Any serious intercurrent or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol including but not limited to:

  * Uncontrolled diabetes mellitus (fasting plasma glucose > 130 mg/dL or 7.2 mmol/L)
  * Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
  * Active infections
  * Gastrointestinal disease limiting the ability to swallow oral medications or absorb oral medications including refractory nausea and vomiting, chronic gastrointestinal diseases, inflammatory bowel disease; malabsorption syndromes
  * Patients with enteric stomata or significant bowel resection
  * Prior history of corneal ulceration
  * Patients with any evidence of severe or uncontrolled systemic liver disease including those with known hepatitis B and hepatitis C (excluding treated hepatitis C that has been cured)
  * Active bleeding diatheses
* Significant active cardiovascular or pulmonary disease including:

  * Uncontrolled hypertension (i.e., systolic blood pressure > 180 mmHg, diastolic blood pressure > 95 mmHg); use of anti-hypertensive agents to control hypertension before cycle 1 day 1 is allowed
  * Pulmonary hypertension
  * Uncontrolled asthma or oxygen (O2) saturation < 90% by arterial blood gas analysis or pulse oximetry on room air
  * Significant valvular disease; severe regurgitation or stenosis by imaging independent of symptom control with medical intervention, or history of valve replacement
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiogram (ECG) e.g. medically significant (symptomatic) bradycardia, complete left bundle branch block, third degree heart block and second-degree heart block or history of arrhythmia requiring an implantable cardiac defibrillator; or within the last 6 months before administration of the first dose of drug:

    * Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation or ventricular tachycardia)
    * Placement of a pacemaker for control of rhythm
    * Ischemic myocardial event, including angina requiring therapy and artery revascularization procedures
    * Ischemic cerebrovascular event, including transient ischemic attack and artery revascularization procedures
    * New York Heart Association (NYHA) class III or IV heart failure
    * Symptomatic pulmonary embolism or asymptomatic pulmonary emboli within the last 3 months
  * Baseline prolongation of the rate-corrected QT interval (QTc) (e.g., repeated demonstration of QTcF >= 470 msec (mean value) obtained from 3 ECGs, using the screening clinic ECG machine derived QTc value, or history of congenital long QT syndrome, or torsades de pointes); any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
  * Left ventricular ejection fraction (LVEF) by either multigated acquisition (MUGA) or echocardiography (ECHO) less than lower limit of normal
* Patients with active malignancies other than NSCLC or prior curatively treated malignancy at high risk of relapse during the study period with the exception of localized squamous or basal cell skin cancers
* Concurrent anti-cancer therapy
* History of hypersensitivity attributed to compounds of similar chemical or biologic composition to MLN0128 (TAK-228) or osimertinib (AZD9291)
* Pregnant women or women who are breast feeding are not eligible for the study; the effects of MLN0128 (TAK-228) and osimertinib (AZD9291) on the developing human fetus are unknown
* Women of non-child bearing potential must be:

  * Women more than 50 years must be post-menopausal for at least 12 months following the end of all exogenous hormonal treatments OR
  * Women under 50 years must be postmenopausal for at least 12 months following the end of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution OR
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
* Women of child bearing potential must have a negative serum or urine pregnancy test within 7 days of registration and must agree to:

  * Practice 1 highly effective method of contraception and 1 additional effective (barrier) method, at the same time, from the time of signing the informed consent through 120 days (or longer, as mandated by local labeling [e.g., United Surgical Partners International (USPI), Summary of Product Characteristics (SmPC), etc.;]) after the last dose of study drug, OR
  * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient; NOTE: Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception; female and male condoms should not be used together
* Male patients, even if surgically sterilized (i.e., status postvasectomy) must agree to:

  * Practice highly effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug, OR
  * Practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient; NOTE: Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner), withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception; female and male condoms should not be used together
  * Not to donate sperm during the course of this study or within 120 days after receiving their last dose of study drug
* Inability to discontinue drugs that are strong cytochrome P450 3A4 (CYP3A4) or P450 3A5 (CYP3A5), cytochrome P450 2C19 (CYP2C19), and cytochrome P450 2C9 (CYP 2C9) inhibitors and/or inducers; and substrates of CYP 3A4/5 or CYP1A2 that are sensitive or have a narrow therapeutic window at least three weeks prior to study registration
* Patients receiving systemic corticosteroids (either IV or oral steroids, excluding inhalers or low-dose hormone replacement therapy) within 1 week before administration of the first dose of study drug
* Consumption of grapefruit or grapefruit juice is not permitted during the study; patients should not consume food or beverages containing the fruit or juice of grapefruits or Seville oranges within 7 days before the first dose of study drug and throughout the study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with MLN0128 (TAK-228) and osimertinib (AZD9291)
* No concomitant use of proton pump inhibitors (PPI) is allowed; any prior PPI must be discontinued at least one week before receiving MLN0128 (TAK-228)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-03-23 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of sapanisertib in combination with osimertinib in patients with EGFRmutant (m) non-small cell lung cancer (NSCLC) | 28 days
  Toxicities will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4 (CTCAE v4). CTCAE version 5.0 will be utilized beginning April 1, 2018.
Dose-limiting toxicity (DLT) of sapanisertib in combination with osimertinib in patients with EGFRm NSCLC | 28 days
  Toxicities will be graded according to the NCI CTCAE v4. CTCAE version 5.0 will be utilized beginning April 1, 2018.

SECONDARY OUTCOMES:
Non-DLTs associated with the administration of sapanisertib and osimertinib | Up to 30 days after completion of study treatment
  Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest. Adverse events will be summarized using all adverse events experienced, although a sub-analysis may be conducted including only those adverse events in which the treating physician deems possibly, probably or definitely attributable to one or both study treatments.
Pharmacokinetic (PK) profiles of sapanisertib in combination with osimertinib | Baseline, and at 1, 2, 4, 6, 8, and 24 hours post-sapanisertib administration, before administration and at 1, 2, 4, 6, 8, and 24 hours post-sapanisertib on day 26 of course 1; and day 1 of course 2
  PK analyses will be descriptive and will permit the evaluation of the PK profile of Tsapanisertib when combined with osimertinib.
Response rate | Up to 2 years
  Will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Summary statistics such as the mean, median, counts and proportion, will be used to describe patients' clinical characteristics. Treatment administered will be reported including the number of cycles, dose modifications, reason off treatment, reason off study, whether a DLT was experienced, best response, and time to progression. These will be listed for each patient and summarized using standard descriptive methods.
Disease control rate | Up to 2 years
  Summary statistics such as the mean, median, counts and proportion, will be used to describe patients' clinical characteristics. Treatment administered will be reported including the number of cycles, dose modifications, reason off treatment, reason off study, whether a DLT was experienced, best response, and time to progression. These will be listed for each patient and summarized using standard descriptive methods.
Progression free survival | From start of treatment to time of progression or death, whichever occurs first, assessed up to 2 years
  Summary statistics such as the mean, median, counts and proportion, will be used to describe patients' clinical characteristics. Treatment administered will be reported including the number of cycles, dose modifications, reason off treatment, reason off study, whether a DLT was experienced, best response, and time to progression. These will be listed for each patient and summarized using standard descriptive methods.
Response rate of patients with T790M- NSCLC in an expansion cohort | Up to 2 years
  Will be assessed using RECIST 1.1. Summary statistics such as the mean, median, counts and proportion, will be used to describe patients' clinical characteristics. Treatment administered will be reported including the number of cycles, dose modifications, reason off treatment, reason off study, whether a DLT was experienced, best response, and time to progression. These will be listed for each patient and summarized using standard descriptive methods.
Disease control rate of patients with T790M- NSCLC in an expansion cohort | Up to 2 years
  Summary statistics such as the mean, median, counts and proportion, will be used to describe patients' clinical characteristics. Treatment administered will be reported including the number of cycles, dose modifications, reason off treatment, reason off study, whether a DLT was experienced, best response, and time to progression. These will be listed for each patient and summarized using standard descriptive methods.
Progression free survival of patients with T790M- NSCLC in an expansion cohort | At 6 months
  Summary statistics such as the mean, median, counts and proportion, will be used to describe patients' clinical characteristics. Treatment administered will be reported including the number of cycles, dose modifications, reason off treatment, reason off study, whether a DLT was experienced, best response, and time to progression. These will be listed for each patient and summarized using standard descriptive methods.
Biomarkers of response and resistance to the combination, explored by studying baseline biopsies, resistance biopsies, and serial plasma deoxyribonucleic acid specimens | Up to 2 years
  Predictors of clinical outcomes will be investigated using logistic regression, Cox proportional hazards regression and or generalized estimating equations as appropriate. Potential predictors include clinical predictors and molecular correlates analyzed in tumor and blood. Descriptive statistics and plotting of data will also be used to better understand potential relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Penelope A Bradbury, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (5):
- United States (3):
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
- Canada (2):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario